CLINICAL TRIAL: NCT03916029
Title: The Hearing for Learning Initiative - a Service-enhancement Model of Ear Health Facilitators to Address the Crisis in Ear and Hearing Health of Aboriginal Children in the Northern Territory: a Stepped-wedge Cluster Randomised Trial
Brief Title: Hearing for Learning Initiative - a Health Facilitator Model for Otitis Media
Acronym: HfLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government); Northern Territory Government of Australia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R813; TEHREC -18-3264 (Other: Ethics Committee); CAHREC - 19-330 (Other: Ethics Committee)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Otitis Media; Conductive Hearing Loss
Keywords: primary health care; workforce; Aboriginal or Torres Strait Islander; facilitator; education
MeSH Terms: conditions — Otitis Media; Hearing Loss, Conductive

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Data analyst will be blinded to the cluster allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Facilitator (Active Comparator): 120 hours training for local community members delivered on-country face-to-face during 6 4-day weeks and over a 3-6 month period. Certificate II modules in Aboriginal Primary Health Care, ear and hearing health skills development (otoscopy, tympanometry, and hearScreen) and employment as Ear Health Facilitators to the end of the trial.
  Interventions: Behavioral: facilitator
- Control (No Intervention): No Facilitator. Brief 6-monthly 2 to 3 hour in-service training via zoom for health professionals.

INTERVENTIONS:
Behavioral: facilitator — Training and employment of community members to assist the diagnosis and management of otitis media
  Arms: Facilitator

SUMMARY:
The Hearing for Learning Initiative is a stepped-wedge cluster randomised controlled trial. The HfLI will implement and rigorously evaluate an innovative community-based service-enhancement model of ear and hearing health, in partnership with participating communities and health and education services.

This initiative will address the following research question: In urban, rural and remote Aboriginal communities in the Northern Territory, does employment, training and integration of local Ear and Hearing Clinical and Education Support Officers into health and education services (the Hearing for Learning initiative), compared to current practice, increase the proportion of children who receive an ear assessment, reduce the prevalence of ear and hearing problems and improve education outcomes of Aboriginal and Torres Strait Islander children, during a four year trial period?

DETAILED DESCRIPTION:
Background: Australian Indigenous children achieve lower scores in school readiness and education outcomes than their non-Indigenous peers. Chronic otitis media and hearing loss during early childhood are associated with lower scores for these outcomes. Local problem: Failure to meet child health program schedules and evidence based practice in ear and hearing health is linked to high turnover of the health workforce, inadequate clinical skills and poor knowledge of ear and hearing health needs of children.

This Hearing for Learning Initiative aims to improve health care and education services.

Interventions: The intervention involves training and employing non-professional community members to facilitate busy primary health care services to deliver evidence-based ear and hearing health assessments in children 0 to 16 years of age, and to facilitate the teaching and home learning of hearing impaired children (the intervention).

Trial design: A stepped-wedge community (n=18) cluster-randomised trial will compare the proportion of children receiving an ear assessment (primary outcomes) in the HfLI (intervention) periods with no HfLI (control) periods. Participating communities will be randomly assigned in 6-monthly steps to shift from control to intervention on pre-specified start dates.

Outcomes: the primary outcome is the change in the proportion of Aboriginal and Torres Strait Islander children who receive an ear assessment, between intervention and control periods.

ELIGIBILITY:
Inclusion Criteria: Aboriginal or Torres Strait Islander, resident in participating community (cluster)

Exclusion Criteria: none

Ages: 1 Week to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-02-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Ear assessment | 6-monthly
  Proportion of children who have had a documented ear assessment

SECONDARY OUTCOMES:
Prevalence of otitis media | 6-monthly
  Proportion of children with any otitis media
Management plan | 6-monthly
  Proportion of otitis media cases with a management plan
Appropriate management plan | 6-monthly
  Proportion of management plans that are appropriate
Follow-up | 6-monthly
  Proportion of cases with follow-up within 10 days

OTHER OUTCOMES:
Prevalence of hearing loss among school age children | 6-monthly
  Proportion of school age children with conductive hearing loss

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Leach, PhD, Principal Investigator — Menzies School of Health Research; Kelvin Kong, MBBS, Study Director — Newcastle University; Peter S Morris, MBBS, PhD, Study Director — Menzies School of Health Research; Alan Cass, MBBS, PhD, Study Director — Menzies School of Health Research
Locations (20):
- Australia (20):
  - Ali Curung, Ali Curung, Northern Territory
  - Ampilatwatja, Ampilatwatja, Northern Territory
  - Darwin, Darwin, Northern Territory
  - Galiwin'ku, Galiwin'ku, Northern Territory
  - Gunbalanya, Gunbalanya, Northern Territory
  - Kalkarindji Primary Health Centre, Kalkarindji, Northern Territory
  - Wurli Wurlinjang Health Service, Katherine, Northern Territory
  - Lajamanu Primary Health Centre, Lajamanu, Northern Territory
  - Mala'la Health Service, Maningrida, Northern Territory
  - Milikapiti Community Health Centre, Milikapiti, Northern Territory
  - Milingimbi Health Clinic, Milingimbi, Northern Territory
  - Minjilang Community Health Centre, Minjilang, Northern Territory
  - Nauiyu, Nauiyu, Northern Territory
  - Palumpa Community Health Centre, Palumpa, Northern Territory
  - Pirlangimpi Health Clinic, Pirlangimpi, Northern Territory
  - Ti Tree Community Health Centre, Ti Tree, Northern Territory
  - Wadeye Community Health Centre, Wadeye, Northern Territory
  - Warruwi Community Health Centre, Warruwi, Northern Territory
  - Julanimawu (Nguiu) Community Health centre, Wurrumiyanga, Northern Territory
  - Yirrkala Clinic, Yirrkala, Northern Territory

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kong K, Cass A, Leach AJ, Morris PS, Kimber A, Su JY, Oguoma VM. A community-based service enhancement model of training and employing Ear Health Facilitators to address the crisis in ear and hearing health of Aboriginal children in the Northern Territory, the Hearing for Learning Initiative (the HfLI): study protocol for a stepped-wedge cluster randomised trial. Trials. 2021 Jun 16;22(1):403. doi: 10.1186/s13063-021-05215-7. PMID 34134736